CLINICAL TRIAL: NCT03699540
Title: Marijuana Effects on Simulated Driving Performance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanna Babalonis, PhD (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Shanna Babalonis, PhD, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 43636; R21DA045101-02 (NIH)
Record Dates: First submitted 2018-10-02; First posted 2018-10-09 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Cannabis; Cannabis Use; Marijuana; Marijuana Usage; Alcohol Drinking
Keywords: simulated driving, outpatient
MeSH Terms: conditions — Marijuana Abuse; Alcohol Drinking | interventions — nabiximols; Ethanol; Exercise

STUDY DESIGN:
Intervention Model Description: Within-subject, randomized, placebo-controlled, double-dummy, double-blind study
Who Masked: Participant, Investigator
Masking Description: Double-blind, double-dummy, placebo-controlled design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Active Marijuana Dose (Experimental): Participants will receive experimental/non-therapeutic dose(s) of active marijuana, under double-blind conditions
  Interventions: Drug: Marijuana
- Inactive Marijuana Dose (Placebo Comparator): Participants will receive experimental/non-therapeutic dose(s) of inactive marijuana, under double-blind conditions
  Interventions: Drug: Inactive marijuana
- Active Alcohol Dose (Active Comparator): Participants will receive experimental/non-therapeutic dose(s) of active alcohol, under double-blind conditions
  Interventions: Drug: Alcohol
- Inactive Alcohol Dose (Placebo Comparator): Participants will receive experimental/non-therapeutic dose(s) of inactive alcohol, under double-blind conditions
  Interventions: Drug: placebo alcohol

INTERVENTIONS:
Drug: Marijuana — Experimental, non-therapeutic administration of active marijuana dose(s)
  Other Names: Active cannabis
  Arms: Active Marijuana Dose
Drug: Alcohol — Experimental, non-therapeutic administration of active alcohol dose(s)
  Other Names: Active alcohol
  Arms: Active Alcohol Dose
Drug: placebo alcohol — Experimental, non-therapeutic administration of inactive alcohol dose(s)
  Arms: Inactive Alcohol Dose
Drug: Inactive marijuana — Experimental, non-therapeutic administration of inactive marijuana dose(s)
  Other Names: inactive cannabis
  Arms: Inactive Marijuana Dose

SUMMARY:
This study will examine the effects of various strains of marijuana on simulated driving performance; the effects of alcohol administration will also be examined to further understand how marijuana-induced driving changes compare to the effects of alcohol. Secondary outcomes will include physiological effects, subjective- and observer-rated outcomes, and psychomotor performance under the various dose conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult participants
* Ages 21-50
* History of marijuana use
* History of alcohol use

Exclusion Criteria:

* Clinically significant medical conditions
* Ongoing/significant drug use outside of marijuana and alcohol use

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data with other outside researchers.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via internet postings (e.g., Craigslist) and locally posted flyers.
Pre-assignment Details: Participants meeting all I/E criteria were invited to enroll. Unique, randomized dose orders were created for each participant. The study utilized a within-subject, randomized, placebo-controlled, double-dummy, double-blind design.
Groups:
- Marijuana Effects on Simulated Driving Performance: Within subject study. Participants will receive experimental/non-therapeutic doses of active/inactive marijuana in combination experimental/non-therapeutic dose of inactive/active alcohol.
Period: Overall Study
Arm/Group | Marijuana Effects on Simulated Driving Performance
Started | 10
Inactive Alcohol/ Tetrahydrocannabinol (THC) 0mg | 8
Inactive Alcohol/THC 15mg | 10
Inactive Alcohol/THC 30mg | 9
Inactive Alcohol/Combined THC 15mg/CBD 7.5mg | 9
Active Alcohol/THC 0mg | 10
Completed | 9
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Completing Participants: Subjects who completed the study
Arm/Group | Completing Participants
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.56 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Peak for Standard Deviation in Lane Position (SDLP)
Description: Standard deviation of lane position (SDLP) of the car is the amount of weaving/swerving of the car in and out of the lane. It is a frequent metric for assessing driving ability.
Time Frame: This outcome was recorded in regular intervals after drug administration for the duration of the session (approx. 9 hrs) and a peak score was calculated across all these time intervals.
Population: Per Protocol population, defined as participants completing the experimental drug conditions.
Measure: Mean (Standard Error); unit: centimeters
Groups:
- Inactive Alcohol / THC 0mg: Participants will receive experimental/non-therapeutic dose of inactive alcohol, under double-blind conditions
  Participants will receive experimental/non-therapeutic dose of inactive marijuana, under double-blind conditions
- Inactive Alcohol / THC 15mg; Inactive Alcohol / THC 30mg: Participants will receive experimental/non-therapeutic dose of inactive alcohol, under double-blind conditions
  Participants will receive experimental/non-therapeutic dose of active marijuana, under double-blind conditions
- Inactive Alcohol / Combined THC 15mg / CBD 7.5mg: Participants will receive experimental/non-therapeutic dose of inactive alcohol, under double-blind conditions
  Participants will receive a combined experimental/non-therapeutic dose of active marijuana and Cannabidiol (CBD), under double-blind conditions
- Active Alcohol / THC 0mg: Participants will receive experimental/non-therapeutic dose of active alcohol, under double-blind conditions
  Participants will receive experimental/non-therapeutic dose of inactive marijuana, under double-blind conditions
Arm/Group | Inactive Alcohol / THC 0mg | Inactive Alcohol / THC 15mg | Inactive Alcohol / THC 30mg | Inactive Alcohol / Combined THC 15mg / CBD 7.5mg | Active Alcohol / THC 0mg
Number analyzed (Participants) | 8 | 9 | 9 | 9 | 9
centimeters | 1.33 (0.09) | 1.37 (0.09) | 1.42 (0.10) | 1.35 (0.08) | 1.77 (0.24)

2. Secondary Outcome: Subject-Rated Outcomes: Mean Peak Score for Driving Difficulty
Description: Participants rated their subjective response on a standardized VAS scale (0 to 100). Higher scores indicate worse outcome/greater impairment. Raw data transformed to peak scores.
Time Frame: This outcome (VAS score) was recorded in regular intervals after drug administration for the duration of the session (approx. 9 hrs) and a peak score was calculated across all these time intervals.
Population: Per Protocol population, defined as participants completing the experimental drug conditions.
Measure: Mean (Standard Error); unit: Score on a scale (0 to 100)
Groups:
- Inactive Alcohol / Combined THC 15mg / CBD 7.5mg: Participants will receive experimental/non-therapeutic dose of inactive alcohol, under double-blind conditions
  Participants will receive a combined experimental/non-therapeutic dose of active marijuana and CBD, under double-blind conditions
Arm/Group | Inactive Alcohol / THC 0mg | Inactive Alcohol / THC 15mg | Inactive Alcohol / THC 30mg | Inactive Alcohol / Combined THC 15mg / CBD 7.5mg | Active Alcohol / THC 0mg
Number analyzed (Participants) | 8 | 9 | 9 | 9 | 9
Score on a scale (0 to 100) | 6.75 (4.46) | 33.89 (10.77) | 40.89 (10.02) | 30.22 (10.10) | 71.89 (9.48)

3. Secondary Outcome: Subject-Rated Outcome: Mean Peak Score for Drug and Alcohol Effect
Description: Participants rated their subjective response on a standardized VAS scale (0 to 100). Higher scores indicate greater drug effects. Raw data transformed to peak scores.
Time Frame: This outcome (VAS scores) was recorded prior to and in regular intervals after drug administration for the duration of the session (approx. 9 hrs)
Population: Per Protocol population, defined as participants completing the experimental drug conditions.
Measure: Mean (Standard Error); unit: Score on a scale (0 to 100)
Arm/Group | Inactive Alcohol / THC 0mg | Inactive Alcohol / THC 15mg | Inactive Alcohol / THC 30mg | Inactive Alcohol / Combined THC 15mg / CBD 7.5mg | Active Alcohol / THC 0mg
Number analyzed (Participants) | 8 | 9 | 9 | 9 | 9
Score on a scale (0 to 100) | 6.13 (2.88) | 32.11 (8.41) | 68.89 (4.66) | 38.44 (8.39) | 71.22 (7.42)

4. Secondary Outcome: Subject-Rated Outcome: Mean Peak Score for Difficulty Concentrating
Description: Participants rated their subjective response on a Likert type scale (Not at all=0, A Little Bit=1, Moderately=2, Quite A Bit=3, Extremely=4). Greater values indicate greater drug effect. Raw data transformed to peak scores.
Time Frame: as for outcome 1
Population: Per Protocol population, defined as participants completing the experimental drug conditions.
Measure: Mean (Standard Error); unit: Score on a scale (0 to 4)
Arm/Group | Inactive Alcohol / THC 0mg | Inactive Alcohol / THC 15mg | Inactive Alcohol / THC 30mg | Inactive Alcohol / Combined THC 15mg / CBD 7.5mg | Active Alcohol / THC 0mg
Number analyzed (Participants) | 8 | 9 | 9 | 9 | 9
Score on a scale (0 to 4) | 0.38 (0.26) | 1.11 (0.26) | 2.22 (0.57) | 0.78 (0.36) | 3.89 (0.95)

5. Secondary Outcome: Observer-Rated Outcome: Mean Peak Score for Relaxed
Description: Research observer rated on a Likert type scale (Not at all=0, A Little Bit=1, Moderately=2, Quite A Bit=3, Extremely=4). Greater values indicate greater drug effect. Raw data transformed to peak scores.
Time Frame: as for outcome 1
Population: Per Protocol population, defined as participants completing the experimental drug conditions.
Measure: Mean (Standard Error); unit: Score on a scale (0 to 4)
Arm/Group | Inactive Alcohol / THC 0mg | Inactive Alcohol / THC 15mg | Inactive Alcohol / THC 30mg | Inactive Alcohol / Combined THC 15mg / CBD 7.5mg | Active Alcohol / THC 0mg
Number analyzed (Participants) | 8 | 9 | 9 | 9 | 9
Score on a scale (0 to 4) | 1.50 (0.19) | 1.67 (0.17) | 2.00 (0.17) | 2.11 (0.11) | 2.11 (0.11)

6. Secondary Outcome: Observer-Rated Outcome: Mean Peak Score for Good Mood
Description: as for outcome 5
Time Frame: as for outcome 1
Population: Per Protocol population, defined as participants completing the experimental drug conditions.
Measure: Mean (Standard Error); unit: Score on a scale (0 to 4)
Arm/Group | Inactive Alcohol / THC 0mg | Inactive Alcohol / THC 15mg | Inactive Alcohol / THC 30mg | Inactive Alcohol / Combined THC 15mg / CBD 7.5mg | Active Alcohol / THC 0mg
Number analyzed (Participants) | 8 | 9 | 9 | 9 | 9
Score on a scale (0 to 4) | 1.25 (0.31) | 1.44 (0.24) | 1.78 (0.15) | 1.89 (0.11) | 2.11 (0.31)

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- Inactive Alcohol / THC 0mgPerformance: Participants will receive experimental/non-therapeutic dose of inactive alcohol, under double-blind conditions Participants will receive experimental/non-therapeutic dose of inactive marijuana, under double-blind conditions
Arm/Group | Inactive Alcohol / THC 0mgPerformance | Inactive Alcohol / THC 15mg | Inactive Alcohol / THC 30mg | Inactive Alcohol / Combined THC 15mg / CBD 7.5mg | Active Alcohol / THC 0mg
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 1/9 | 1/9 | 2/9 | 1/9 | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inactive Alcohol / THC 0mgPerformance (N=9) | Inactive Alcohol / THC 15mg (N=9) | Inactive Alcohol / THC 30mg (N=9) | Inactive Alcohol / Combined THC 15mg / CBD 7.5mg (N=9) | Active Alcohol / THC 0mg (N=9)
stomachache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Chills (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Muscle/limb pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2023-12-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT03699540/Prot_ICF_001.pdf
  • Statistical Analysis Plan (2023-12-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT03699540/SAP_002.pdf